CLINICAL TRIAL: NCT04437199
Title: A 12-Week, Double-blind, Randomised, Placebo-controlled, Parallel Group Study to Investigate the Efficacy and Safety of Daily Administration of Tricaprilin as AC-SD-03 in Participants With Migraine
Brief Title: Tricaprilin Phase 2 Pilot Study in Migraine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cerecin (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AC-20-022
Record Dates: First submitted 2020-06-11; First posted 2020-06-18 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — tricaprylin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AC-SD-03 (Active Comparator): Tricaprilin SD formulation, twice daily. Administered orally
  Interventions: Drug: Tricaprilin
- AC-SD-03P (Placebo Comparator): Placebo formulation, twice daily. Administered orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tricaprilin — Powder formulation will be mixed with 240 mL water and shaken until fully dispersed.
  Each dosing unit of 12.5 g of AC-SD-03 contains 5 g of the active ingredients (tricaprilin)
  Other Names: AC-SD-03
  Arms: AC-SD-03
Drug: Placebo — Powder formulation will be mixed with 240 mL water and shaken until fully dispersed.
  Other Names: AC-SD-03P
  Arms: AC-SD-03P

SUMMARY:
This is a randomised, double-blind, placebo-controlled, parallel-group, multi-centre study of tricaprilin as AC-SD-03 compared with placebo for the reduction of migraine in participants with frequent migraine.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be 18 to 70 years of age inclusive, at the time of signing the informed consent.
2. Participants who have frequent (episodic or chronic) migraine with or without aura, for at least 1 year, according to the International Classification of Headache Disorders version 3 beta (ICHD 3-beta), age at time of onset must be <50 years.
3. Participants must have a certain number of migraine headaches days per month, as confirmed by the baseline measurement period.
4. Use of one allowed migraine prophylactic is permitted if the participant has been on a stable dose for at least 2 months prior to the screening.
5. Participants must have failed (no therapeutic response) 1-4 migraine prophylactic treatments.
6. The participant is able to tolerate a 12.5g dose of AC-SD-03 (containing 5g of tricaprilin) as per sentinel dose challenge at the Baseline Visit.
7. From Visit 2 to Visit 3 (baseline measurement period), the participant has sufficient compliance (at least 80%) with daily eDiary headache entries.

Exclusion Criteria:

1. In the opinion of the Investigator, has presence or history of an advanced, severe, progressive, or unstable disease of any type that could interfere with efficacy and safety assessments, or put the participant at risk.
2. Use of barbiturates (and/or butalbital-containing analgesics) or opioids (and/or opioid-containing analgesics) for migraine acute treatment ≥ 4 days per month on average and/or in the last month prior to Screening Visit.
3. Use in the last 3 months prior to Screening Visit of CGRP agents, Botox injections, TENS, cranial nerve blocks, trigger-point injections, acupuncture, CBD-containing products, infusion therapy.
4. Current use, or use within 3 months of Visit 2 (baseline), of Axona® or other MCT-containing products (such as coconut oil). Use of MCT-containing products is not allowed at any time during trial participation.
5. Current use, or use within 3 months prior to Screening, of a ketogenic diet, low-carb diet, intermittent fasting (including the 5:2 diet). Ketogenic diets, low-carb diet, intermittent fasting (including the 5:2 diet) are not allowed during the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2022-02-07 (Actual); Study Completion 2022-02-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the number of migraine headache days during Month 3 (ΔMDMth3) | 12 weeks
  Number of migraine headache days using headache diary parameters

SECONDARY OUTCOMES:
Change from baseline in the number of migraine headache days during Month 1 (ΔMDMth1) and Month 2 (ΔMDMth2) of treatment and overall, from Months 1-3 | 4, 8, 12 weeks
  Number of migraine headache days using headache diary parameters
The proportion of participants with a 50% reduction from baseline in number of migraine headache days in treatment months 1, 2, and 3 | 4, 8, 12 weeks
  Response rate defined as a reduction in number of migraine headache days
Change from baseline in monthly acute migraine medicine use during treatment months 1, 2 and 3 | 4, 8, 12 weeks
  Acute migraine medicine use during treatment
Change from baseline Headache Impact Test (HIT-6) score at the end of Months 1, 2 and 3 | 4, 8, 12 weeks
  Headache Impact Test (HIT-6) score. Total score range between 36-78 (higher score indicates a worse impact)

OTHER OUTCOMES:
Change from baseline in the number of headache days (migraine and non-migraine headache) during treatment months 1, 2 and 3 (ΔHDMth1, ΔHDMth2 and ΔHDMth3) | 4, 8, 12 weeks
  Headache diary parameters
Change from baseline in MIDAS score at the end of Month 1, 2 and 3 | 4, 8, 12 weeks
  Migraine Disability Assessment Scale (MIDAS) score. Total score range between 0-28 (higher score indicates more severe disability)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Cerecin
Locations (10):
- Australia (10):
  - Paratus Clinical Central Coast, Kanwal, New South Wales
  - Holdsworth House, Sydney, New South Wales
  - Calvary Adelaide Hospital, Adelaide
  - Paratus Clinical Research Western Sydney, Blacktown
  - Paratus Clinical Research Brisbane, Brisbane
  - Emeritus Research, Camberwell
  - Paratus Clinical Research Canberra, Canberra
  - Austin Health Hospital, Heidelberg
  - Alfred Health Hospital, Melbourne
  - Gold Coast University Hospital, Southport

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chow L, Presanis J, McIntyre N, Henderson S, Bloch M, Hutton E, Cantillon M. Tricaprilin (CER-0001) for the preventive treatment of migraine: A phase 2 randomised, double-blind, placebo-controlled pilot study. J Neurol Sci. 2024 Sep 15;464:123147. doi: 10.1016/j.jns.2024.123147. Epub 2024 Jul 22. PMID 39094432